CLINICAL TRIAL: NCT06337292
Title: Incisional Negative Pressure Wound Therapy to Reduce Infection and Complications in High-Risk Fractures: A Multicenter Randomized Controlled Trial
Brief Title: Incisional Negative Pressure Wound Therapy to Reduce Infection and Complications in High-Risk Fractures
Acronym: iVAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00440042
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Fracture of Tibia; Wound Heal; Infected Wound; Wound Complication; Wound Dehiscence
MeSH Terms: conditions — Tibial Fractures; Wound Infection

STUDY DESIGN:
Intervention Model Description: Randomization into study treatment arms (incisional NPWT or non-suction standard of care) will occur in variable permuted blocks, stratified by clinical center, in a 1:1 ratio. Patients will be randomized electronically by an online Data Management System maintained by the Coordinating Center at Johns Hopkins School of Public Health.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Wound Care (No Intervention): Patients randomized to the control group will receive standard wound care.
- Incisional Negative Pressure Wound Therapy (NPWT) (Experimental): Patients randomized to the treatment group will receive wound care which includes the application of an incisional negative pressure wound vacuum.
  Interventions: Device: Incisional Negative Pressure Wound Therapy (NPWT)

INTERVENTIONS:
Device: Incisional Negative Pressure Wound Therapy (NPWT) — Participants in the treatment group will be standardized and will receive incisional NPWT using the any incisional VAC system that can apply 75-125mmHg continuous suction to the incision. The VAC sponge will be placed over the surgical wound at least 2cm in width and >3cm in length.
  Arms: Incisional Negative Pressure Wound Therapy (NPWT)

SUMMARY:
This is a multi-center, pragmatic, parallel arm randomized controlled trial (RCT) of 352 patients with high-risk open or closed tibial plateau fracture, high-risk open or closed tibial pilon fracture, or open tibial shaft fracture with incision >3cm. Eligible participants will be randomized to receive either incisional negative pressure wound therapy (NPWT) or a non-suction standard-of-care wound dressing for their definitive wound management. The primary outcome will be a composite outcome to evaluate clinical status 3 months after randomization. The secondary outcomes will independently assess the components of the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. All open or closed tibial plateau or pilon fractures treated operatively with internal fixation at high risk for complication. Any open Gustilo Type I, II or IIIA tibial shaft fracture treated definitively with internal or external fixation with or without ipsilateral leg compartment syndrome if at least one wound is primarily closed.
2. We define high-risk fractures as those that are either:

   * Closed fracture initially treated with an external fixator (with or without limited internal fixation) and treated definitive more than 3 days later after swelling has resolved;
   * Any open type I, II or IIIA fracture, regardless of timing of definitive treatment;
   * Any tibial plateau fracture associated with ipsilateral leg compartment syndrome fasciotomy wounds that has at least one wound primarily closed
3. Requiring incision for fixation or debridement of 3 cm or greater.
4. Patients 18 years of age or older

Exclusion Criteria:

1. The study injury is already infected at time of study enrollment.
2. Patient is unable to receive incisional NPWT for any reason.
3. Patients who have already had definitive fixation prior to enrollment in the study.
4. Severe problems with maintaining follow-up (e.g., patients who are homeless at the time of injury or those who are intellectually challenged without adequate family support or who are prisoners).
5. The study injury is a Gustilo Type IIIB or IIIC open fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complication composite outcome | 3 months
  The primary outcome will be a composite outcome. We will hierarchically assess the components of the composite outcome in the following order: (1) all-cause mortality, (2) injury-related amputation of the lower extremity, (3) number of surgeries to treat a deep or organ space infection (CDC criteria), (4) wound healing complications requiring reoperation, (5) nonoperative wound necrosis at 2 or 6 weeks, wound dehiscence at 2 or 6 weeks or superficial infection (CDC criteria), (6) SCAR-Q Symptom Scale, (7) SCAR-Q Appearance Scale

CONTACTS AND LOCATIONS:
Overall Officials: I. Leah Gitajn, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Renan Castillor, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - University of Maryland R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire

IPD SHARING:
Plan to Share IPD: No